CLINICAL TRIAL: NCT02684890
Title: Detection of Emotions in a Spoken Language Among Tinnitus Patients
Acronym: EMSLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Oron Yahav, ENT Specialist, Wolfson Medical Center
Other Study IDs: 0220-15-WOMC
Record Dates: First submitted 2016-02-13; First posted 2016-02-18 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tinnitus patients: Patients with tinnitus lasting over 3 months
- Non-tinnitus patients: Patients without tinnitus

SUMMARY:
Tinnitus may affect the ability of patients to detect emotions in spoken language. This study will compare this ability between tinnitus patients and non-tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus lasting 3 months and longer
* Hebrew speakers

Exclusion Criteria:

* Tinnitus which began less than 3 months ago Learned Hebrew after the age of 5

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with tinnitus
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Emotion scores | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Centre, Holon, Israel

IPD SHARING:
Plan to Share IPD: No